CLINICAL TRIAL: NCT05247957
Title: NKG2D CAR-NK Cell Therapy in Patients With Relapsed or Refractory Acute Myeloid Leukemia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: end
Sponsor: Hangzhou Cheetah Cell Therapeutics Co., Ltd (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CARNK-001
Record Dates: First submitted 2022-01-20; First posted 2022-02-21 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Safety and Efficacy
Keywords: NKG2D CAR-NK; Relapsed or Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Recurrence; Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NKG2DL-specific CAR-NK cells (Experimental): Experimental: NKG2DL-specific CAR-NK cells, 2 infusions on Day 0 and Day 7 After preconditioning with chemotherapy, NKG2DL-specific CAR-NK cells will be evaluated
  Interventions: Biological: CAR-NK cells

INTERVENTIONS:
Biological: CAR-NK cells — NKG2DL-specific CAR-NK cells, 2 infusions on Day 0 and Day 7
  Other Names: NKG2DL-specific CAR-NK cells

SUMMARY:
This trial will explore the maximum tolerated dose of cord blood NKG2D CAR-NK in the treatment of recurrent refractory acute myeloid leukemia in a dose-escalation manner, and observe its clinical safety and efficacy.

DETAILED DESCRIPTION:
This is a single arm, open-label, Phase 1 study initiated with 3 cohorts:

Cohort 1: 2×10∧6/kg CAR-NK cells, 2 infusions on Day 0 and Day 7 Cohort 2: 6×10∧6/kg CAR-NK cells, 2 infusions on Day 0 and Day 7 Cohort 3: 18×10∧6/kg CAR-NK cells, 2 infusions on Day 0 and Day 7

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥ 10 years old and ≤ 75 years old, male or female;
2. Meet the diagnostic criteria for recurrent AML: detection of leukemia cells after complete remission (CR) or >0.1% of leukemia cells in bone marrow, including recurrence after allogeneic hematopoietic stem cell transplantation, or extramedullary infiltration of leukemia cells;
3. Initial cases with failure of 2 lines of standard treatment; patients who relapsed within 12 months after consolidation intensification after CR; recurrence in 12 months and no respond to conventional chemotherapy; 2 or more recurrences; persistent extramedullarial leukemia;
4. Patients currently have no effective treatment options, such as chemotherapy or allogeneic hematopoietic stem cell transplantation, or patients voluntarily choose to infuse NKG2D CAR-NK cells as the first treatment option;
5. Physical status assessment (ECOG-PS) of the Eastern Oncology Collaborative Group is 0-2 points;
6. Estimated survival > 3 months
7. Flow cytometry check for NKG2D ligand expression on the surface of cancer cells for a reference of selecting patients
8. The main organs of the patient are well functioned: (1) cardiac function: no heart disease or coronary heart disease, the patient's cardiac function grade 1-2; (2) liver function: TBIL≦3ULN, AST≦2.5ULN, ALT≦2.5ULN; (3) Renal function: Cr≦1.25ULN;
9. The patient's peripheral superficial vein can meet the needs of intravenous injection;
10. No other serious diseases that conflict with this protocol (e.g., autoimmune diseases, immunodeficiency, organ transplantation);
11. No history of other malignant tumors;
12. Women of childbearing age must be tested negative for pregnancy within 7 days, and subjects of childbearing age must use appropriate contraception during both the trial and for 3 months after the test;
13. Subjects have negative HIV, HBV, HCV, syphilis serology test results
14. Written informed consent form must be signed before enrollment.

Exclusion Criteria:

1. Acute promyelocytic leukemia (type M3);
2. Patients with cardiac insufficiency, patients with hepatic and renal insufficiency;
3. Those who need treatment with other malignant tumors;
4. Poorly controlled hypertension (systolic blood pressure >160 mmHg and/or diastolic blood pressure >90 mmHg) or clinically significant cardiovascular and cerebrovascular diseases such as cerebrovascular accident (within 6 months before signing the informed consent form), myocardial infarction (within 6 months before signing the informed consent), unstable angina, congestive heart failure, or severe arrhythmias that cannot be controlled with drugs or have a potential impact on research treatment;
5. Also suffering from other hematologic diseases (such as hemophilia, myelofibrosis, etc., which researchers consider unsuitable for inductees);
6. Diffuse vascular internal coagulation;
7. Concomitant serious infection or other serious underlying medical condition;
8. Have immunodeficiency and autoimmune diseases;
9. Have severe allergic diseases;
10. Clinical symptoms of brain dysfunction or severe mental illness that can not understand or follow the research protocol;
11. Have participated in clinical trials of other drugs within 4 weeks or within 21 days of surgery;
12. Have received cell therapy in the previous 1 month;
13. Have received hormonal drug therapy in the previous 14 days;
14. Known HIV-positive patients or hepatitis B and C patients and syphilis patients;
15. Have received organ transplants (excluding stem cell transplant patients);
16. Drug abuse, medical, psychological or social conditions that may interfere with a subject's participation in the study or evaluation of the results of the study;
17. Pregnant or lactating women;
18. Those who cannot be followed up as scheduled;
19. Investigator considers that the subject has any clinical or laboratory abnormalities or compliance problems and is not suitable to participate in this clinical study.

Ages: 10 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-10-13 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity | 28 days
  To evaluate the clinical safety and short-term efficacy of NKG2D ligand-specific umbilical cord blood CAR-NK cells in the treatment of patients with relapsed refractory acute myeloid leukemia by intravenous infusion
Maximal Tolerable Dose | 28 days
  tolerability evaluationtransplantation after intravenous infusion of NKG2D ligand-specific umbilical cord blood CAR-NK cells for patients with relapsed refractory acute myeloid leukemia

SECONDARY OUTCOMES:
leukemia-free survival#LFS# | 52weeks
  leukemia-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Peihua Lu, MD, Principal Investigator — Hebei Yanda Lu Daopei Hospital
Locations (1):
- Hebei Yanda Lu Daopei Hospital, Sanhe, Hebei, China

IPD SHARING:
Plan to Share IPD: No